CLINICAL TRIAL: NCT07245823
Title: Randomized Study Evaluating the Treatment of Vulvovaginal Gaping by Plication of the Puborectalis Muscles Versus Perineorrhaphy ± Transverse Myorrhaphy of the Puborectalis Muscles at 12 Months.
Brief Title: Randomized Study Evaluating the Treatment of Vulvovaginal Gaping by Plication of the Puborectalis Muscles Versus Perineorrhaphy ± Transverse Myorrhaphy of the Puborectalis Muscles at 12 Months. (HERA)
Acronym: HERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A01362-45
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prolapse Genital; Vulvovaginal Disease
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sagittal plication of the puborectal muscles reconstruction (Experimental): Anatomical reconstruction of the vulvovaginal gape by sagittal plication of the puborectal muscles
  Interventions: Procedure: Anatomical reconstruction of the vulvovaginal gape; Other: Questionnaires; Radiation: MRI
- Perineorrhaphy ± transverse myorrhaphy of the puborectal muscles reconstruction (Active Comparator): Anatomical reconstruction of the vulvovaginal gape by perineorrhaphy ± transverse myorrhaphy of the puborectal muscles
  Interventions: Procedure: Anatomical reconstruction of the vulvovaginal gape; Other: Questionnaires; Radiation: MRI

INTERVENTIONS:
Procedure: Anatomical reconstruction of the vulvovaginal gape — Anatomical reconstruction of the vulvovaginal gape with two different surgeries
Other: Questionnaires — Questionnaires of quality of sexual life (PPSSQ), of anal incontinence and constipation
Radiation: MRI — MRI of the genital hiatus

SUMMARY:
Vulvovaginal incompetence is generally associated with prolapse and contributes to the pathogenesis of the latter. The perineum and the perineal body (PB) are structures frequently injured throughout life, leading to vesicourethral and rectoanal dysfunction, which are the main focus of study. Other symptoms, such as periorificial dyspareunia and vulvovaginal incompetence, appear to be less verbalized by women. The resulting sexual discomfort is linked, on the one hand, to physical anatomical trauma, with, in some cases, vulvovaginal incompetence contributing to a vaginal sensitivity decreased, and, on the other hand, to psychological trauma with damage to self-image. Vulvoperineoplasty is a surgical repair procedure that aims to optimally reconstruct the introital anatomy by correcting the vulvovaginal incompetence in order to restore normal anatomy, restore self-image, and treat the symptoms of vaginal laxity (feeling of a vagina that is too large and loss of vaginal sensitivity).

Conventional surgical techniques for treating vulvar incompetence, such as levator myorrhaphy and perineorrhaphy, are currently being questioned because they cause functional sequelae, particularly regarding to sexual quality of life. The pubo-rectal muscle plication (PPR) technique is based on the anatomical observation of puborectalis muscle lengthening (PMR) observed on MRI scans in patients with vaginal incompetence. This technique could be an interesting alternative in the surgical treatment of vulvovaginal incompetence.

The main objective of this study is to evaluate the effectiveness of anatomical reconstruction of vulvovaginal incompetence by sagittal plication of the puborectalis muscles vs. by perineorrhaphy ± transverse myorrhaphy of the puborectalis muscles at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Female patient between 18 and 80 years-old.
* Genital hiatus at rest ≥ 4 cm by POP-Q
* Sexually active woman without pain (never/rarely scored) during penetration and who has stopped sexual activity due to vulvovaginal incompetence without pain (never/rarely scored) during penetration
* Prolapse
* Candidate for surgery for anatomical reconstruction of the vulvovaginal incompetence
* Patient affiliated with a social security scheme or beneficiary of such a scheme, according to Article L.1124-1 of the Public Health Code
* Free, informed and signed consent

Exclusion Criteria:

* Resting GH < 4 cm (POP-Q classification)
* Women not sexually active and not planning to become sexually active
* Chronic perineal pain syndrome
* Anal sphincter injury with concomitant indication for sphincterorrhaphy
* Cognitive or language impairment of the patient unable to complete the study questionnaires
* Contraindications to surgery or anesthesia
* Adult under guardianship, curatorship, or other legal protection, deprived of liberty by judicial or administrative decision, hospitalized without consent
* Pregnant, breastfeeding, or parturient woman
* Patient planning to become pregnant during the study period
* Immediate postpartum

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2029-04-20 (Estimated); Study Completion 2029-04-25 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of anatomical reconstruction of vulvovaginal gaping | 12 months
  The effectiveness of anatomical reconstruction of the vulvovaginal gap will be assessed at 12 months using a composite criterion. The reconstruction will be considered successful if the following three criteria are met:
  * Resting GH < 4 cm,
  * AND PGI-I "overall condition" improved or greatly improved,
  * AND pain during intercourse rated "never or rarely" (question 6 of the PPSSQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Dijon Bourgogne, Dijon, France